CLINICAL TRIAL: NCT00518674
Title: Local Anesthetics After Total Knee Arthroplasty: Intra- vs. Extraarticular Administration? A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Local Anesthetics After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KF01329190
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-07

CONDITIONS: Postoperative Pain
Keywords: pain; local infiltration analgesia
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: local infiltration analgesia — local wound infiltration with 30 ml ropivacaine 0.2 % (60 mg)

SUMMARY:
The aim of this randomized, double-blind and placebo-controlled study is to evaluate the specific role of injection of local anesthetic into the intra- vs. extraarticular tissues after toal knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed oral and written consent to participate
* Able to speak Danish

Exclusion Criteria:

* Treatment with opioids
* Body Mass Index > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale pain score

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Andersen, MD, Principal Investigator — Hvidovre University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen LO, Kristensen BB, Madsen JL, Otte KS, Husted H, Kehlet H. Wound spread of radiolabeled saline with multi- versus few-hole catheters. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):200-2. doi: 10.1097/aap.0b013e3181c7733d. PMID 20301825